CLINICAL TRIAL: NCT02921204
Title: Study is to Assess the Effect of Dietary Intake of Nutrients and Level of Vitamin D in Women
Brief Title: Dietary Intake and Vitamin D Level in Adult Women
Acronym: VDAW
Status: Completed | Type: Observational
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Collaborators: University of Connecticut (Other)
Responsible Party: Principal Investigator, Nora ALfaris, Profossor, Princess Nourah Bint Abdulrahman University
Other Study IDs: NON
Record Dates: First submitted 2016-09-29; First posted 2016-10-03 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Deficiency of Vitamin D3
Keywords: Vitamin D; Calcium; Phytic Acid; body weight
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Vitamin D status: Subjects are recruited to asses Vitamin D status with no interventions
  Interventions: Other: Vitamin D status

INTERVENTIONS:
Other: Vitamin D status — There is no intervention in this study

SUMMARY:
Vitamin D deficiency is most diagnosed among women living in the Kingdom of Saudi Arabia. Many factors have been attributed to the incidence of vitamin D deficiency. Saudi women are thought to be at greater risk for vitamin D deficiency because of their darker skin type and the likelihood of reduced ultraviolet exposure . The present study entitled, "Dietary Intake and Vitamin D Level in adult Women," was formulated as there is paucity of data on the etiologic importance of dietary intake in Vitamin D level on blood on women. The major objective of the proposed study is to assess the effect of dietary intake of nutrients and level of vitamin D in women .

DETAILED DESCRIPTION:
For this study, the investigators enrolled 168 women 35-55 years old to evaluate Vitamin D status and to determined whether status was correlated with Vitamin D deficiency.

All women completed a self-administered questionnaire about personal socio-demographic characteristics; They all had anthropometric measurements of body mass index and waist circumference. A 24-hour dietary recall was administered to all women.

The proximate analysis of 25 types of food was conducted according to the American Association of Organic Chemists (AOAC) methods. The following parameters were measured: serum calcium. Vitamin D, levels of parathyroid hormone.

ELIGIBILITY:
Inclusion Criteria:

* Women 35- 55 years old,
* Women who spoke Arabic language fluently, and
* Women who were willing to fill a 24-hour questionnaire and provide a serum sample for measurements.

Exclusion Criteria:

* Women < 35 years old or > 55 years old.

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pre and post-menopausal women 35-55 years of age who were able to provide a 24 hour dietary record.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Vitamin D serum levels | 1 year

SECONDARY OUTCOMES:
Calcium serum levels | 1 year
Vitamin D and Calcium Intake | 1 year

OTHER OUTCOMES:
Exposure to sun | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Amani Aljajani, PhD, Study Chair — Princess Nourah Bint Abdulrahman University

IPD SHARING:
Plan to Share IPD: Undecided